CLINICAL TRIAL: NCT05353699
Title: Implementation of a Comprehensive Intervention on Hypertension（HTN） and Type 2 Diabetes Mellitus（DM） at PHC Level: a Hybrid Type II Cluster-controlled Multisite Effectiveness-implementation Trial
Brief Title: Implementation of a Comprehensive Intervention on Hypertension（HTN） and Type 2 Diabetes Mellitus（DM） at PHC Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Center for Chronic and Noncommunicable Disease Control and Prevention, China CDC (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Shiqihu
Record Dates: First submitted 2022-02-28; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention groups (Experimental)
  Interventions: Other: Implementation strategies
- Control groups (No Intervention): as same as before

INTERVENTIONS:
Other: Implementation strategies — We will adopt implementation strategies,which include Capacity-building strategies, Supervision, Integration strategies, Implementation process strategies, Dissemination strategies, Scale-up strategies.Firstly,Capacity-building strategies include:recruit, designate, and train for leadership; work with educational institutions.Secondly,Supervision includes provide clinical supervision;Thirdly,Integration strategies include: remind clinicians; use data warehousing techniques.Fourthly,Implementation process strategies include: identify and prepare champions; identify early adopters; inform local opinion leaders; involve patients/consumers and family members; obtain and use patients/consumers and family feedback.Fifthly,Dissemination strategies include: make training dynamic.Finally,Scale-up strategies include: use train-the-trainer strategies;place innovation on fee for service lists/formularies.
  Arms: Intervention groups

SUMMARY:
Background: The disease burden of hypertension(HTN) and type 2 diabetes mellitus(DM) is rising rapidly in China.Comprehensive interventions(Implementation strategies for providers and interventions for patients) are critical to strengthen primary health care systems and address the burden of multiple comorbidities. In order to promote equal access to health services and narrow the gap in population health, China has launched the national Essential Public Health Services Equity Programme (EPHSEP) nationwide. EPHSEP contains guidelines for health management services for HTN and type 2 DM. The program has been in operation for 10 years. However, the management of HTN and type 2 DM in China is far from satisfactory. The purpose of this study is to understand current control and management situation of HTN and type 2 DM, investigate the barriers and facilitators in the implementation of HTN and type 2 DM service delivery standards, propose feasible implementation strategies,implement in certain areas,and to evaluate the effectiveness of interventions and the performance and impact of implementation strategies.

Methods: Based on previous work,four community health service centres and four township health centres will be selected in West Coast District of Qingdao city of Shandong province,Suzhou City of Jiangsu province, Changsha city of Hunan province and Luohe city of Henan Province.In each of the four provinces,one community health service center and one township health center will be selected.Two community health service centres and two township health centres will be selected as the intervention groups, and the other community health service centres and township health centres will be selected as the control groups.

The study will be divided into three phases: Phase 1, 2 and 3. Phase 1 and phase 2 cross-sectional studies are the basis for phase 3 intervention studies.

Phase 1 will be conducted from March 2022 to April 2022.In phase 1, a quantitative questionnaire survey will be conducted among 5464 HTN and 7040 type 2 DM patients in 8 community health service centers to obtain the data of awareness rate, screening rate, diagnosis rate, treatment rate, control rate and management service of hypertension and type 2 diabetes patients,so as to understand current control and management situation of HTN and type 2 DM.

Phase 2 will be conducted in April 2022. In phase 2, about 64 medical staff and related managers providing HTN and type 2 DM health management services and 80 patients with HTN and type 2 DM in 8 community health service centers will be investigated through qualitative interviews,so as to investigate the barriers and facilitators in the implementation of HTN and type 2 DM service delivery standards and to propose feasible implementation strategies.

Phase 3 will be conducted a mixed-methods type 2 hybrid effectiveness-implementation study from May 2022 to January 2023. Interventions are divided into four levels through a cascading model of screening, diagnosis, treatment, and control. Implementation strategies are divided into 6 categories according to Implementation Mapping: Capacity-building strategies（Recruit, designate, and train for leadership; Work with educational institutions), Supervision(Provide clinical supervision), Integration strategies(Remind clinicians; Use data warehousing techniques), Implementation process Strategies(Identify and prepare champions; Identify early adopters; Inform local opinion leaders; Involve patients/consumers and family members; Obtain and use patients/consumers and family feedback), Dissemination strategies(Make training dynamic), Scale-up strategies(Use train-the-trainer strategies;Place innovation on fee for service lists/formularies). We will adopt between site design to select 4（2*2 ）community health service centers and 4（2*2）township health centers, among which 2 community health service centers and 2 township health centers will implement the strategy, while the other selected sites will not implement the strategy. The 2*2 community health service centers and 2*2 township health centers will be divided into group matching control and self pre- and post-control. In phase 3, 2280 patients with HTN and 2656 patients with type 2 DM will be surveyed by quantitative questionnaire, and about 64 medical staff and related managers providing HTN and type 2 DM health management services will be surveyed by qualitative interview. This is to implement improved implementation strategies and to assess the effectiveness of interventions and the performance and impact of implementation strategies.

ELIGIBILITY:
For the quantitative questionnaire survey, the demander's population in phase 1 will include a total of 5464 patients with HTN and 7040 patients with type 2 DM in the 8 selected primary medical institutions.The demander's population in phase 2 is the same as that in phase 1.In phase 3, the demander's population will include a total of 2280 patients with HTN and 2656 patients with type 2 DM in the 8 selected primary medical institutions.

* Inclusion criteria for respondents:①Patients with HTN and type 2 DM who have received basic public health service management for more than one year, and have no plan to move within the next year; ②Have normal communication ability and independent behavior ability; ③Volunteer to participate in the project questionnaire survey and provide the informed consents.
* Exclusion criteria for respondents:①Patients with severe chronic diseases or in acute stage who cannot cooperate with investigators; ②Mental disorders or cognitive disorders (including dementia, cognitive impairment, deafness, etc.).

For the qualitative interview component, the provider's population will include policy-decision makers, managers, health professionals, healthcare workers who provide health management services for HTN and type 2 DM, and stakeholders who contain governmental officials/staff from civil society/non-governmental organization.Focus group discussions (FGDs) will be conducted. At each level, a group of people gets together for focus groups.During the interview, the specific number of interviewees shall be determined according to the principle of information saturation.

* Inclusion criteria for interviewees:①Health care personnel responsible for community HTN or type 2 DM management; ②Responsible for the national basic public health service project -HTN, type 2 DM health management work for at least 12 months; ③Willing to participate in the project; ④Willing to be interviewed;⑤Good presentation and verbal communication skills.
* Exclusion criteria for interviewees:①Health care workers who were not responsible for hypertensive or diabetic management;②Health care workers who carried out the management for less than 12 months;③Those who are not willing to participate in the project;④Unwilling to be interviewed;⑤Lack of expressive ability or difficulty in communicating in Mandarin; The demander's population will include a total of 80 patients with HTN and type 2 DM in the selected 8 primary medical institutions. The qualitative interview mainly adopts the personal in-depth interview method to understand the main problems in the implementation of the intervention measures, explore the causes of the problems, and possible improvement measures and suggestions.
* Inclusion criteria include:①patients who have participated in management;②patients who are active in conversation;③patients who are willing to participate in interviews.
* Exclusion criteria for patients:①patients with hypertension or diabetes who do not participate in the management;②patients who are not willing to be interviewed.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12648 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Awareness change：Change from Baseline Awareness at 3, 6,9 months | during the intervention; immediately after the intervention
  Awareness of HTN/ type 2 DM in population:% awareness towards HTN/ type 2 DM in population.Survey method will be used to assess this outcome measure.
Screening rate change：Change from Baseline Screening rate at 3, 6,9 months | during the intervention; immediately after the intervention
  Screening rate of patients with HTN/ type 2 DM:% patients with HTN/ type 2 DM screened among those who have ever screened blood pressure/blood sugar.Data will be obtained from administrative record.
Diagnostic rate change：Change from Baseline Diagnostic rate at 3, 6,9 months | during the intervention; immediately after the intervention
  Diagnostic rate of patients with HTN/ type 2 DM:% patients with HTN/ type 2 DM diagnosed among those who have been screened blood pressure/blood sugar.Data will be obtained from administrative record.
Treatment rate change：Change from Baseline Treatment rate at 3, 6,9 months | during the intervention; immediately after the intervention
  Treatment rate of patients with HTN:% patients with HTN who took antihypertensive drugs in the last two weeks was determined among those who have been diagnosed blood pressure; Treatment rate of patients with type 2 DM:% patients with type 2 DM who have taken treatment measures (including lifestyle intervention and/or medication) among those who have been diagnosed blood sugar.Data will be obtained from administrative record.
Control rate change：Change from Baseline Control rate at 3, 6,9 months | during the intervention; immediately after the intervention
  Control rate of patients with HTN/type 2 DM:% patients whose blood pressure/ blood sugar are controlled among those who have been treated.Data will be obtained from administrative record.
Implementation strategies use change: Change from Baseline Implementation at 3, 6,9 months | during the intervention; immediately after the intervention
  Implementation strategies use:qualitative interviews with managers of health centers.Interviews method will be used to assess this outcome measure.
Supervision change: Change from Baseline Implementation at 3, 6,9 months | during the intervention; immediately after the intervention
  Supervision model: % scheduled supervision field visits completed.Data will be obtained from administrative data.
Referral completeness change: Change from Baseline Implementation at 3, 6,9 months | during the intervention; immediately after the intervention
  Referral completeness: % referrals completed as prescribed by the clinical algorithm.Data will be obtained from administrative data.
Adaptations to protocol change: Change from Baseline Implementation at 3, 6,9 months | during the intervention; immediately after the intervention
  Adaptations to protocol during intervention period: qualitative interviews with managers of local health department and health centers.Interviews method will be used to assess this outcome measure.
Implementation change: Change from Baseline Implementation at 3, 6,9 months | during the intervention; immediately after the intervention
  Qualitative assessment: qualitative interviews with managers of health.Interviews method will be used to assess this outcome measure.

SECONDARY OUTCOMES:
Coverage change: Change from Baseline Reach at 3, 6,9 months | during the intervention; immediately after the intervention
  Coverage of population receiving health service for HTN and type 2 DM:proportion of target population receiving HTN and DM service.Data will be obtained from administrative data.
Screening coverage of eligible for HTN change: Change from Baseline Reach at 3, 6,9 months | during the intervention; immediately after the intervention
  Screening coverage of eligible for HTN:proportion of eligible for HTN receiving screening.Data will be obtained from administrative data.
Screening coverage of eligible for type 2 DM change: Change from Baseline Reach at 3, 6,9 months | during the intervention; immediately after the intervention
  Screening coverage of eligible for type 2 DM:proportion of eligible for type 2 DM receiving screening.Data will be obtained from administrative data.
Coverage of screening for patients with HTN/type 2 DM change: Change from Baseline Reach at 3, 6,9 months | during the intervention; immediately after the intervention
  Coverage of screening for patients with HTN/type 2 DM:% patients with HTN/type 2 DM who have been screened for hypertension/ diabetes.Data will be obtained from administrative data.
Readiness change: Change from Baseline Adoption at 3, 6,9 months | during the intervention; immediately after the intervention
  Readiness for implementation:a checklist to check readiness for implementation using.Data will be obtained from administrative data.
Health centers/clinic's adoption change: Change from Baseline Adoption at 3, 6,9 months | during the intervention; immediately after the intervention
  Health centers/clinic's adoption: % proportion of health centers/clinics implemented lifestyle intervention and/or medication.Data will be obtained from administrative data.
PHC professional's adoption change: Change from Baseline Adoption at 3, 6, 9 months | during the intervention; immediately after the intervention
  PHC professional's adoption:% of PHC professionals trained in implementing the guidelines for HTN and DM.Data will be obtained from administrative data.
Timely adoption | during the intervention
  Timely adoption：# early adopters at the local site. Observation methods will be used to assess this outcome measure.
Leader adoption change: Change from Baseline Adoption at 3, 6,9 months | during the intervention; immediately after the intervention
  Leader adoption: # leaders recruited/designated/trained for the change effort in intervention implementation.Interview and observation methods will be used to assess this outcome measure.
Institution adoption change: Change from Baseline Adoption at 3, 6,9 months | during the intervention; immediately after the intervention
  Institution adoption:% intended Institution incorporated Administrative of HTN and DM in their routine service systems.Interview and observation methods will be used to assess this outcome measure.
Follow-up fidelity change: Change from Baseline Fidelity at at 3, 6,9 months | during the intervention; immediately after the intervention
  Follow-up fidelity: % patients with "adequate" number of follow-up visits received.Data will be obtained from administrative data(records).
Health professionals implemented guidelines/protocol change: Change from Baseline Fidelity at at 3, 6,9 months | during the intervention; immediately after the intervention
  Health professionals implemented guidelines /protocol: % of PHC professionals implemented according to the guidelines/protocol in actual work. Interview and observation methods will be used to assess this outcome measure.
Qualitative assessment-Behavior changes sustained (staff) | 15 months
  Long-term maintenance of changes in management behavior related to hypertension/type 2 DM. Interview and observation methods will be used to assess this outcome measure.
HTN and type 2 DM institutionalized | immediately after the intervention
  HTN and type 2 DM become institutionalized or part of the routine organizational practices.Data will be obtained from administrative data and survey.
Settings continue the intervention | immediately after the intervention
  proportion and representativeness of settings that continue the intervention.Data will be obtained from administrative data.
Total intervention cost | immediately after the intervention
  Total intervention cost per patient.Data will be obtained from administrative data.
Total treatment cost | immediately after the intervention
  Total treatment cost per patient.Data will be obtained from administrative data.
Intervention maintenance costs | immediately after the intervention
  % breakdown of maintenance (recurring) costs (ongoing training, personnel, materials, and other).Data will be obtained from administrative data.
Facility vs. community costs | immediately after the intervention
  % of costs of healthcare divided between facility level and community level.Data will be obtained from administrative data.
out-of-pocket patient costs | immediately after the intervention
  % out-of-pocket patient costs.Survey method will be used to assess this outcome measure.
Qualitative assessment-maintenance: | immediately after the intervention
  Interviews method will be used to assess this outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- National Center for Chronic and Noncommunicable Disease Control and Prevention, Chinese Center for Disease Control and Prevention, Beijing, Beijing Municipality, China